CLINICAL TRIAL: NCT02047201
Title: Assessing Tumor Response and IMRT Treatment Planning After Induction Chemotherapy Based on FDG-PET/CT for Locally Advanced Head and Neck Squamous Cell Carcinoma.
Brief Title: Assessing Tumor Response and IMRT Treat Plan After IC Based on FDG-PET/CT for Locally Advanced HNSCC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Lithuanian University of Health Sciences (Other)
Responsible Party: Principal Investigator, Ilona Kulakiene, Professor, Lithuanian University of Health Sciences
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EHNCTE-1309
Record Dates: First submitted 2014-01-22; First posted 2014-01-28 (Estimated); Last update posted 2016-03-02 (Estimated); Status verified 2016-03

CONDITIONS: Head and Neck Squamous Cell Carcinoma
Keywords: Head and neck cancer; PET/CT; induction chemotherapy; IMRT
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Head and Neck Neoplasms | interventions — Radiotherapy, Intensity-Modulated; Docetaxel; Fluorouracil; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Experimental (Experimental): Induction chemotherapy (Docetaxel, Cisplatin and Fluorouracil) following radiochemotherapy (IMRT using PET/CT images after IC for treatment planning + cisplatin iv 40 mg/m2 weekly).
  Interventions: Radiation: IMRT; Radiation: PET/CT; Drug: Docetaxel; Drug: Fluorouracil; Drug: Cisplatin

INTERVENTIONS:
Radiation: IMRT — IMRT treatment planning using FDG-PET/CT images after induction chemotherapy (IC).
  Other Names: intensity-modulated radiation therapy
Radiation: PET/CT — Assessing tumor response using FDG-PET/CT.
  Other Names: Positron emission tomography-computed tomography
Drug: Docetaxel — 75 mg/m2, IV (in the vein) on day 1 every 3 weeks. Number of cycles: 3.
  Other Names: Taxotere, Docefrez
Drug: Fluorouracil — 750 mg/m2 continuous infusion for 120 h IV (in the vein) every 3 weeks. Number of cycles: 3.
  Other Names: 5-Fluorouracil, Adrucil
Drug: Cisplatin — 75 mg/m2, IV (in the vein) on day 1 every 3 weeks. Number of cycles: 3.
  Other Names: Platinol

SUMMARY:
To evaluate the safety and efficacy of cisplatin plus intensity-modulated radiotherapy (IMRT) based on FDG-PET/CT after induction chemotherapy (IC) for locally advanced head and neck squamous cell carcinoma.

DETAILED DESCRIPTION:
Current guidelines define that pre-IC target volumes must be used for radiotherapy (RT) planning. This prospective, phase II trial assessed the results of patients with locally advanced squamous cell carcinoma of head and neck treatment with IC following by chemoradiotherapy (CRT), using post-IC PET/CT images for IMRT planning.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients aged 18 years or over;
* Histologically confirmed locally advanced (stage III and IV) head and neck squamous cell carcinoma (HNSCC);
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1;
* Signed written informed consent approved by the Lithuanian Bioethics Committee (LBEC);

Exclusion Criteria:

* Positive serum pregnancy test in women of childbearing potential or breastfeeding;
* Presence of distant metastasis;
* Second primary tumor;
* History of other malignancy within the last 5 years;
* Recurrent head and neck cancer;
* Serious uncontrolled concomitant disease that would contraindicate the use of any drugs use in this study as chemotherapy or radiotherapy; ;
* Inadequate organ function, evidenced by the following laboratory results:

  1. Absolute neutrophil count <1,500 cells/mm3;
  2. Platelet count <100,000 cells/mm3;
  3. Hemoglobin <9 g/dL;
  4. Total bilirubin greater than the upper limit of normal (ULN);
  5. AST (SGOT) or ALT (SGPT) >1,5 x ULN;
  6. Alkaline phosphatase levels >2,5 x the ULN;
  7. Serum creatinine >2,0 mg/dl or 177 umol/l.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2013-06; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Progression free survival (PFS) | 24 months after treatment
  PFS was defined as the time from the first day of IC first cycles to either progression or death.

SECONDARY OUTCOMES:
Tumour metabolic response (MTV) reduction (%) | 2 weeks after IC
  MTV was defined as the tumor volume with FDG uptake segmented by a gradient-based method and fixed threshold methods at >40% of SUVmax. The MTV predictive value for tumor response to IC was assessed by comparing MTV's reduction (MTV of second PET/CT difference from MTV of first PET/CT in percent) in IC responders versus non responders and correlation with PFS and OS.
Total lesion glycolysis (TLG) reduction (%) | 2 weeks after IC
  The TLG was defined as (MTV) x (SUVmean). The TLG predictive value for tumor response to IC was assessed by comparing TLG reduction (TLG of second PET/CT difference from TLG of first PET/CT in percent) in IC responders versus non responders and correlation with PFS and OS.
SUVmax reductions (%) | 2 weeks after IC
  The SUVmax was defined as (tissue activity) (mcCi/ml)/(injected dose) (mCI)/(patient weight) (kg) within the voxel having the highest activity within a given region of interest (ROI). The SUVmax predictive value for tumor response to IC was assessed by comparing reductions in SUVmax (SUVmax of second PET/CT difference from SUVmax of first PET/CT in percent) in IC responders versus non responders and correlation with PFS and OS.
Number (%) of participants with adverse events | 12 and 24 months from chemoradiotherapy
  Treatment acute toxicity during IC and CRT (chemoradiotherapy) was weekly assessed according to the National Cancer Institute Common Toxicity Criteria (NCI CTCAE) v.4.0. Late adverse events related with radiotherapy were assessed every three months after CRT using RTOG (Radiation Therapy Oncology Group) /EORTC (European Organization for Research and Treatment of Cancer) toxicity criteria.
Overall survival (OS) | 24 months after treatment
  OS was defined as the time from the first day of IC first cycles until death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Ilona Kulakiene, Prof., Principal Investigator — Lithuanian University of Health Sciences
Locations (1):
- Lithuanian University of Health Sciences, Kaunas, Lithuania

IPD SHARING:
Plan to Share IPD: Yes
3-7/07/2016 in ASCO (American Society of Clinical Oncology) Annual Meeting, Chicago